CLINICAL TRIAL: NCT00336609
Title: Risk and Outcomes of Mucositis in Subjects Being Treated for Breast, Colorectal, Head and Neck, Non-Small Cell Lung Cancers or Non-Hodgkin's Lymphoma
Brief Title: TRIAD Burden of Illness Mucositis Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TRIAD Burden of Illness (Other)
Other Study IDs: No. 200509024
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Gastrointestinal Mucositis (Defined as Mucositis Involving the Mouth, Esophagus, or Small Intestine)
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Observational (non-drug) study to look at the risks and burden of mucositis (sores) involving the mouth, throat and intestines in patients receiving chemotherapy and radiation therapy treatment for various cancer types.

DETAILED DESCRIPTION:
This comprehensive, observational study will prospectively elicit the true incidence (risk) and health and economic burdens of mucosal toxicities associated with anti-cancer drug and radiation therapy. This study will examine the burden of illness of gastrointestinal mucositis (defined as mucositis involving the mouth, esophagus, or small intestine) in the most significant regimens used to treat the most common types of cancers. It is an international investigation in which 1600 patients being treated with specific regimens for cancers of the head and neck, breast, colon, lung (NSCLC)and Non-Hogkin's Lymphoma will be prospectively enrolled from centers throughout the US, Canada, Europe and Australia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Ability to understand the protocol and willing to provide written informed consent
* Membership in one of the following sub-cohorts:

  1. Histologically proven oral cavity or oropharyngeal cancers planned to receive a full cycle of daily single fraction radiation therapy (with or without boost) or IMRT +/- chemotherapy.
  2. Histologically proven laryngeal or hypopharyngeal cancers planned to receive a full cycle of daily single fraction radiation (with or without boost) +/- chemotherapy.
  3. Histologically proven adenocarcinoma of the colon or rectum planned to receive a minimum of 2 cycles of FOLFOX +/- Avastin or Erbitux.1 cycle defined as 2 doses of FOLFOX.
  4. Histologically proven adenocarcinoma of the colon or rectum planned to receive a minimum of 2 cycles of FOLFIRI +/- Avastin or Erbitux. 1 cycle defined as 2 doses of FOLFIRI.
  5. Adenocarcinoma of the breast planned to receive a minimum of 2 cycles of TAC.
  6. Histologically proven adenocarcinoma (any primary) planned to receive a minimum of 2 cycles of capecitabine.
  7. Adenocarcinoma of the breast planned to receive standard or dose-dense doxorubicin and cyclophosphamide (AC) followed by paclitaxel (T) (4 cycles AC followed by 2 cycles T).
  8. Stage 3A or 3B non-small cell lung cancers planned to receive daily single fraction radiation with or without boost (1 fraction daily for 5-6 weeks) +/- Carbo/Taxol.
  9. B-cell Non-Hodgkin's lymphoma (NHL) planned to receive at least 2 cycles of CHOP-14, CHOEP-14, CHOP-DI-14, EPOCH-14 or CHOP-21 +/- rituxan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600
Dates: Start 2005-11; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Sonis T Sonis, DMD, DMSc, Principal Investigator — Brigham and Women's Hospital; Dorothy Keefe, MD, Principal Investigator — University of Adelaide; Linda Elting, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Univeristy Of Wisconsin, Madison, Wisconsin, United States